CLINICAL TRIAL: NCT03334695
Title: An Exploratory, Phase 2a, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Prophylactic Efficacy of a Single Immunization of Ad26.RSV.preF Against Respiratory Syncytial Virus Infection in a Virus Challenge Model in Healthy 18 to 50 Year-Old Adults
Brief Title: An Exploratory Study to Evaluate the Prophylactic Efficacy of a Single Immunization of Ad26.RSV.preF Against Respiratory Syncytial Virus Infection in a Virus Challenge Model in Healthy 18 to 50 Year-old Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Vaccines & Prevention B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CR108398; 2017-003194-33 (EudraCT Number); VAC18193RSV2002 (Other: Janssen Vaccines & Prevention B.V.)
Record Dates: First submitted 2017-10-16; First posted 2017-11-07 (Actual); Results first posted 2021-07-23 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group 1: Ad26.RSV.preF (Experimental): Participants will receive single intramuscular injection of 1*10^11 virus particles (vp) of Ad26.RSV.preF during Day -90 to Day -28. On Day 0, intranasal challenge with respiratory syncytial virus (RSV)-A Memphis 37b virus will occur for all participants.
  Interventions: Biological: Ad26.RSV.preF
- Group 2: Placebo (Placebo Comparator): Participants will receive single intramuscular injection of placebo as sterile 0.9 percent (%) saline for injection during Day -90 to Day -28. On Day 0, intranasal challenge with RSV-A Memphis 37b virus will occur for all participants.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Ad26.RSV.preF — Ad26.RSV.preF will be administered as intramuscular injection at a dose of 1*10^11 vp in single-use vials.
  Other Names: JNJ-64400141
  Arms: Group 1: Ad26.RSV.preF
Drug: Placebo — Placebo will be administered as sterile 0.9% saline for injection.
  Arms: Group 2: Placebo

SUMMARY:
The purpose of this study is to assess a trend for the prophylactic efficacy of a single dose of 1*10^11 virus particles (vp) of adenovirus serotype 26 respiratory syncytial virus pre-fusion F protein (Ad26.RSV.preF) administered intramuscularly to adults aged 18-50 years in the respiratory syncytial virus (RSV) challenge model in terms of reduction of nasal wash viral load compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Each participant must sign an Informed Consent Form (ICF) indicating that he or she understands the purpose of and procedures required for the study, is willing to participate in the study and attend all scheduled visits, is willing to be isolated and stay in the clinic for the quarantine phase, and is willing and able to comply with all study procedures and adhere to the prohibitions and restrictions specified in this protocol
* Participants must be in good health, without significant medical illness, on the basis of a medical evaluation that reveals the absence of any clinically relevant abnormality and includes a physical examination (including height and weight), skin examination, medical history, vital signs (systolic and diastolic blood pressure and heart rate, respiratory rate, and body temperature), and the results of clinical laboratory tests performed within 56 days of vaccination. If there are abnormalities, the participant may be included only if the investigator judges the abnormalities or deviations from normal to be not clinically significant. This determination must be recorded in the participant's source documents and initialed by the investigator
* Participants must have a non-clinically significant 12-lead electrocardiogram (ECG) within 56 days of vaccination including: normal sinus rhythm (heart rate between 50 and 100 beats per minute [bpm], extremes included); QT interval corrected for heart rate according to Fridericia (QTcF) interval less than or equal to (<=) 450 millisecond (ms); QT interval corrected for heart rate according to Bazett (QTcB) interval <= 450 ms; QRS interval less than (<) 120 ms; PR interval <= 210 ms
* Participants must be sero-suitable for respiratory syncytial virus (RSV) within 90 days of vaccination (low immunity to the RSV-A Memphis 37b virus using a virus neutralization assay
* Participant must be healthy on the basis of clinical laboratory tests performed within 56 days of vaccination. If the results of the laboratory screening tests are outside the local laboratory normal reference ranges and additionally within the limits of toxicity Grade 1 according to the US Food and Drug Administration (FDA) toxicity tables (that is, for tests in the FDA table), the participant may be included only if the investigator judges the abnormalities or deviations from normal to be not clinically significant and appropriate and reasonable for the population under study. This determination must be recorded in the participant's source documents and initialed by the investigator

Exclusion Criteria:

* Participant has acute illness (this does not include minor illnesses such as diarrhea) or temperature greater than or equal to (>=) 37.8 degree Centigrade within 24 hours prior to study vaccination
* Participant has history of malignancy (exceptions are basal cell carcinomas of the skin treated over 5 years prior to vaccination considered cured with minimal risk of recurrence)
* Participant has chronic active hepatitis B or hepatitis C infection, documented by hepatitis B surface antigen and hepatitis C antibody, respectively

Viral Challenge Exclusion Criteria:

* Participants having donated or lost more than 1 unit of blood (470 milliliter [mL]) within 60 days or more than one unit of plasma within 7 days
* Participants with active acute respiratory infection

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2017-10-16 (Actual); Primary Completion 2018-07-10 (Actual); Study Completion 2018-11-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Vaccines & Prevention B.V. Clinical Trial, Study Director — Janssen Vaccines & Prevention B.V.
Locations (1):
- hVIVO Services Limited, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In total, 64 participants were screened. Of these, 63 participants were randomized and received the study vaccine. One participant was randomized in error and did not receive the study vaccine hence not included in the analyses.
Groups:
- Ad26.RSV.preF (1*10^11 vp): Participants received a single intramuscular injection of 1*10^11 vp (viral particles) of adenovirus serotype 26 respiratory syncytial virus pre-fusion conformation-stabilized F protein (Ad26.RSV.preF) on Day -28 followed by intranasal challenge with a respiratory syncytial virus (RSV)-A Memphis 37b virus on Day 0 (24 to 90 days after vaccination).
- Placebo: Participants received a single intramuscular injection of matching placebo on Day -28 followed by intranasal challenge with RSV-A Memphis 37b virus on Day 0 (24 to 90 days after vaccination).
Period: Overall Study
Arm/Group | Ad26.RSV.preF (1*10^11 vp) | Placebo
Started | 31 | 32
Completed | 27 | 26
Not Completed | 4 | 6
Not completed — Lost to Follow-up | 3 | 3
Not completed — Physician Decision | 1 | 2
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ad26.RSV.preF (1*10^11 vp) | Placebo | Total
Number analyzed (Participants) | 31 | 32 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.9 (6.19) | 25.9 (6.56) | 25.9 (6.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 6 | 18
  Male | 19 | 26 | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 30 | 32 | 62
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 24 | 28 | 52
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 2 | 3 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  UNITED KINGDOM | 31 | 32 | 63

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Viral Load-Time Curve (VL-AUC) of Respiratory Syncytial Virus (RSV) by Quantitative Reverse Transcriptase-Polymerase Chain Reaction (qRT-PCR)
Description: VL-AUC for RSV was determined by qRT-PCR assay of nasal wash samples. Here, values below the lower limit of quantification (LLOQ) were imputed with zero.
Time Frame: From Day 2 to Day 12
Population: The Intent-to-treat-Challenge (ITTc) population is a subset of the Full Analysis Set (FAS) (all participants who were randomized and received study vaccine, regardless of the occurrence of protocol deviations) included all randomized, vaccinated and challenged participants.
Measure: Median (Inter-Quartile Range); unit: log10 copies*hour per millilitre (h/mL)
Arm/Group | Ad26.RSV.preF (1*10^11 vp) | Placebo
Number analyzed (Participants) | 27 | 26
log10 copies*hour per millilitre (h/mL) | 0 [0.0 to 268.8] | 236 [20.3 to 605.8]
Statistical Analysis 1: Comparison: Ad26.RSV.preF (1*10^11 vp) vs Placebo; Test type: Superiority; p = 0.012, Wilcoxon Rank Sum test

2. Secondary Outcome: Peak Viral Load of RSV-A Memphis 37b
Description: Peak viral load of RSV-A Memphis 37b was defined as the maximum viral load as determined by quantitative RT-PCR assay of nasal wash samples. Here, values below the lower limit of quantification (LLOQ) were imputed with zero.
Time Frame: From Day 2 to Day 12
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: log10 copies per mL
Arm/Group | Ad26.RSV.preF (1*10^11 vp) | Placebo
Number analyzed (Participants) | 27 | 26
log10 copies per mL | 0.000 [0.000 to 4.539] | 5.365 [3.027 to 6.665]

3. Secondary Outcome: Viral Load by Quantitative RT-PCR Assay on Day 6 and 7
Description: Viral load determined by quantitative RT-PCR assay of nasal wash samples on Day 6 and Day 7 were reported. Here, values below the lower limit of quantification (LLOQ) were imputed with zero.
Time Frame: Day 6 (0 hour and 12 hours) and Day 7 (0 hour and 12 hours)
Population: The Intent-to-treat-Challenge (ITTc) population is a subset of the Full Analysis Set (FAS) (all participants who were randomized and received study vaccine, regardless of the occurrence of protocol deviations) included all randomized, vaccinated and challenged participants. Here 'n' (number analyzed) signifies the number of participants analyzed for this outcome measure (OM) at specified timepoints.
Measure: Mean (Standard Error); unit: log10 copies per mL
Arm/Group | Ad26.RSV.preF (1*10^11 vp) | Placebo
Number analyzed (Participants) | 27 | 26
log10 copies per mL
  Day 6: 0 hour | 0.821 (0.349) | 2.898 (0.630)
  Day 6: 12 hour: number analyzed (Participants) | 26 | 26
  Day 6: 12 hour | 1.261 (0.433) | 2.939 (0.604)
  Day 7: 0 hour | 1.761 (0.436) | 3.072 (0.586)
  Day 7: 12 hour: number analyzed (Participants) | 27 | 25
  Day 7: 12 hour | 1.552 (0.443) | 3.025 (0.530)

4. Secondary Outcome: VL-AUC of RSV by Quantitative Culture of RSV (Plaque Assay) on Day 6 and 7
Description: VL-AUC of RSV by the quantitative culture of nasal wash samples on Day 6 and Day 7 were determined.
  pfu*h/mL stands for plaque-forming units hour per millilitre.
Time Frame: Day 6 (0 hour and 12 hours) and Day 7 (0 hour and 12 hours)
Population: The Intent-to-treat-Challenge (ITTc) population is a subset of the Full Analysis Set (FAS) (all participants who were randomized and received study vaccine, regardless of the occurrence of protocol deviations) included all randomized, vaccinated and challenged participants. Here 'n' (number analyzed) signifies the number of participants analyzed for this OM at specified timepoints.
Measure: Mean (Standard Error); unit: log10 pfu*h/mL
Arm/Group | Ad26.RSV.preF (1*10^11 vp) | Placebo
Number analyzed (Participants) | 27 | 26
log10 pfu*h/mL
  Day 6: 0 hour | 0.278 (0.1936) | 1.587 (0.4159)
  Day 6: 12 hour | 0.304 (0.2198) | 1.737 (0.4320)
  Day 7: 0 hour | 0.101 (0.1015) | 1.226 (0.3505)
  Day 7: 12 hour: number analyzed (Participants) | 27 | 25
  Day 7: 12 hour | 0.276 (0.1931) | 1.237 (0.3891)

5. Secondary Outcome: Percentage of Participants With Symptomatic RSV Infections
Description: Symptomatic RSV infection is defined in two ways (Conservative and Liberal). Conservative: participant had 2 or more quantifiable RT-PCR measurements on different samples, with one of following: symptoms of 2 different categories of subject symptom card (SSC) (Upper Respiratory [runny/stuffy nose, sneezing, sore throat, earache], Lower Respiratory [cough, shortness of breath, chest tightness, wheeze], Systemic [malaise, headache, muscle and/or joint ache]) regardless of grade and assessment timepoint or Grade 2 symptom from any category; Liberal (RT-PCR): had 2/more quantifiable RT-PCR measurements, with clinical symptom of any severity.
Time Frame: From Day 2 to Day 12
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Ad26.RSV.preF (1*10^11 vp) | Placebo
Number analyzed (Participants) | 27 | 26
Percentage of participants
  Conservative | 22.2 | 46.2
  Liberal | 33.3 | 61.5

6. Secondary Outcome: Total Clinical Symptoms Score at Day 6 and 7
Description: The total clinical symptom score was determined as the sum of the scores (grades) ranges from 0 (no symptom) to 52 (severe symptoms) of the 13 self-reportable symptoms on the SSC. Clinical symptoms includes runny nose, stuffy nose, sneezing, sore throat, ear ache, malaise, headache, muscle and/or joint ache, chilliness/ feverishness, cough, chest tightness, shortness of breath and wheeze. For every separate symptom, the score ranges from 0 (I have no symptom) to 4 (its quite bothersome most of the times and stop from participating in activities).
Time Frame: Day 6 and 7: morning, afternoon and evening
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Ad26.RSV.preF (1*10^11 vp) | Placebo
Number analyzed (Participants) | 27 | 26
Units on a scale
  Day 6: Morning | 0.6 (0.18) | 2.6 (0.64)
  Day 6: Afternoon | 0.4 (0.18) | 2.8 (0.74)
  Day 6: Evening | 0.5 (0.28) | 2.5 (0.65)
  Day 7: Morning | 0.6 (0.23) | 2.5 (0.70)
  Day 7: Afternoon | 0.6 (0.32) | 2.5 (0.70)
  Day 7: Evening | 0.6 (0.32) | 2.5 (0.63)

7. Secondary Outcome: Weight of Mucus Secretions Over Time
Description: The weight mucous over time was determined in grams using eCRF forms. Participants were given pre-weighed packets of paper tissues. After each tissue was used for nose blowing or sneezing, the participants should store them in an airtight plastic bag to calculate the weight of mucus from Day 0 to Day 12. All paper tissues used by each participant were collected for each 24-hour period up to Day 12, to determine daily mucus weight.
Time Frame: Day 0, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11 and 12
Population: as for outcome 4
Measure: Mean (Standard Error); unit: Grams
Arm/Group | Ad26.RSV.preF (1*10^11 vp) | Placebo
Number analyzed (Participants) | 27 | 26
Grams
  Day 0: number analyzed (Participants) | 27 | 25
  Day 0 | 0.586 (0.1883) | 0.175 (0.0913)
  Day 1: number analyzed (Participants) | 26 | 25
  Day 1 | 0.228 (0.0621) | 0.086 (0.0333)
  Day 2: number analyzed (Participants) | 27 | 25
  Day 2 | 0.997 (0.2350) | 0.428 (0.1459)
  Day 3: number analyzed (Participants) | 27 | 25
  Day 3 | 0.970 (0.2176) | 0.543 (0.1333)
  Day 4 | 1.164 (0.3535) | 0.714 (0.2123)
  Day 5 | 1.440 (0.8609) | 1.068 (0.3539)
  Day 6 | 1.226 (0.4925) | 3.132 (1.0991)
  Day 7 | 1.715 (0.7201) | 5.124 (1.3257)
  Day 8 | 0.799 (0.2960) | 3.230 (1.1022)
  Day 9 | 1.004 (0.4147) | 1.798 (0.4406)
  Day 10 | 0.907 (0.3457) | 1.785 (0.4838)
  Day 11 | 0.749 (0.2430) | 1.172 (0.3442)
  Day 12 | 0.622 (0.2647) | 0.990 (0.3005)

8. Secondary Outcome: Number of Tissues Used Over Time
Description: Number of tissues used by participant per time point were reported using eCRF forms. Participants were given pre-weighed packets of paper tissues. After each tissue was used for nose blowing or sneezing, the participants should store them in an airtight plastic bag to calculate the number of tissues used from Day 0 to Day 12. All paper tissues used by each participant were collected for each 24-hour period up to Day 12, to determine daily number of tissues used.
Time Frame: Day 0, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11 and 12
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Tissues
Arm/Group | Ad26.RSV.preF (1*10^11 vp) | Placebo
Number analyzed (Participants) | 27 | 26
Tissues
  Day 0 | 1.8 (0.53) | 0.7 (0.33)
  Day 1 | 1.7 (0.41) | 0.7 (0.27)
  Day 2 | 2.9 (0.65) | 1.2 (0.32)
  Day 3 | 1.9 (0.45) | 1.3 (0.28)
  Day 4 | 2.3 (0.49) | 1.5 (0.31)
  Day 5 | 2.1 (0.81) | 2.3 (0.68)
  Day 6 | 2.4 (0.77) | 5.1 (1.59)
  Day 7 | 2.8 (0.92) | 8.1 (1.94)
  Day 8 | 2.0 (0.71) | 5.2 (1.38)
  Day 9 | 2.3 (0.72) | 2.8 (0.53)
  Day 10 | 1.8 (0.61) | 2.7 (0.61)
  Day 11 | 1.6 (0.47) | 2.0 (0.50)
  Day 12 | 1.4 (0.40) | 1.7 (0.45)

9. Secondary Outcome: Percentage of Participants With Unsolicited Adverse Events (AEs)
Description: Unsolicited AEs are all AEs for which participants were specifically not questioned in the participant diary. An AE is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with a clear causal relationship with the relevant investigational product.
Time Frame: Up to 28 days post-vaccination and up to 28 days post-challenge
Population: The Full Analysis Set (FAS) included all participants who were randomized and received at least one dose of study vaccine, regardless of the occurrence of protocol deviations. Here 'n' (number analyzed) included all evaluable participants who were analyzed at specified categories.
Measure: Number; unit: Percentage of participants
Arm/Group | Ad26.RSV.preF (1*10^11 vp) | Placebo
Number analyzed (Participants) | 31 | 32
Percentage of participants
  Post-vaccination | 35.5 | 46.9
  Post-challenge: number analyzed (Participants) | 27 | 26
  Post-challenge | 74.1 | 69.2

10. Secondary Outcome: Percentage of Participants With Serious Adverse Events (SAEs)
Description: A SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: Up to 6 months post-vaccination and up to 6 months post-challenge
Population: as for outcome 9
Measure: Number; unit: Percentage of participants
Arm/Group | Ad26.RSV.preF (1*10^11 vp) | Placebo
Number analyzed (Participants) | 31 | 32
Percentage of participants
  Post-vaccination | 0 | 0
  Post-challenge: number analyzed (Participants) | 27 | 26
  Post-challenge | 3.2 | 0

11. Secondary Outcome: Percentage of Participants With Solicited Local and Systemic AEs
Description: Solicited local AEs: erythema, swelling/induration, and pain/tenderness. Solicited systemic AEs: fatigue, headache, myalgia, arthralgia, chills, nausea and fever.
Time Frame: 7 days post-vaccination (Day -21)
Population: The Full Analysis Set (FAS) included all participants who were randomized and received at least one dose of study vaccine, regardless of the occurrence of protocol deviations.
Measure: Number; unit: Percentage of participants
Arm/Group | Ad26.RSV.preF (1*10^11 vp) | Placebo
Number analyzed (Participants) | 31 | 32
Percentage of participants
  Solicited local AEs | 100.0 | 18.8
  Solicited systemic AEs | 100.0 | 50.0

12. Secondary Outcome: Percentage of Participants With Vital Signs Abnormalities
Description: Percentage of participants with vital signs abnormalities were reported. Vital signs measurements included body temperature (measured in degree celsius from less than [<] 37.5 to <39.5), respiratory rate, systolic and diastolic blood pressure, and pulse rate, which were graded by FDA Toxicity Grading Scale Grade 0 (=no grade), Grade 1 (=mild), Grade 2 (=moderate), Grade 3 (=severe) and Grade 4 (=potentially life-threatening).
Time Frame: Up to Day 28 post-challenge
Population: as for outcome 9
Measure: Number; unit: Percentage of participants
Arm/Group | Ad26.RSV.preF (1*10^11 vp) | Placebo
Number analyzed (Participants) | 31 | 32
Percentage of participants
  Post-dose: Temperature (<37.5) | 64.5 | 93.8
  Post-dose: Temperature (37.5-<38.0) | 22.6 | 3.1
  Post-dose: Temperature (38.0-<38.5) | 6.5 | 0
  Post-dose: Temperature (38.5-<39.0) | 6.5 | 3.1
  Post-dose: Bradycardia (pulse): Grade 1 | 12.9 | 3.1
  Post-dose: Bradycardia (pulse): Grade 2 | 6.5 | 6.3
  Post-dose: Bradycardia (pulse): Grade 3/4 | 3.2 | 0
  Post-dose: Hypertension (diastolic): Grade 1 | 0 | 3.1
  Post-dose: Hypertension (diastolic): Grade 2 | 6.5 | 0
  Post-dose: Hypertension (systolic): Grade 1 | 3.2 | 3.1
  Post-dose: Respiratory rate: Grade 1 | 25.8 | 18.8
  Post-dose: Tachycardia (pulse): Grade 1 | 3.2 | 0
  Post-challenge: Bradycardia (pulse): Grade 1: number analyzed (Participants) | 27 | 26
  Post-challenge: Bradycardia (pulse): Grade 1 | 18.5 | 11.5
  Post-challenge: Bradycardia (pulse): Grade 2: number analyzed (Participants) | 27 | 26
  Post-challenge: Bradycardia (pulse): Grade 2 | 3.7 | 3.8
  Post-challenge: Bradycardia (pulse): Grade 3/4: number analyzed (Participants) | 27 | 26
  Post-challenge: Bradycardia (pulse): Grade 3/4 | 3.7 | 0
  Post-challenge: Hypertension (diastolic): Grade 1: number analyzed (Participants) | 27 | 26
  Post-challenge: Hypertension (diastolic): Grade 1 | 3.7 | 0
  Post-challenge: Hypertension (systolic): Grade 1: number analyzed (Participants) | 27 | 26
  Post-challenge: Hypertension (systolic): Grade 1 | 0 | 7.7
  Post-challenge: Respiratory rate: Grade 1: number analyzed (Participants) | 27 | 26
  Post-challenge: Respiratory rate: Grade 1 | 25.9 | 26.9
  Post-challenge: Tachycardia (pulse): Grade 1: number analyzed (Participants) | 27 | 26
  Post-challenge: Tachycardia (pulse): Grade 1 | 3.7 | 0

13. Secondary Outcome: Percentage of Participants With Electrocardiogram (ECG) Abnormalities
Description: ECG parameters included heart rate, PR, QRS, QTcB, QTcF, and the uncorrected QT interval which were graded by FDA Toxicity Grading Scale Grade 0 (=no grade), Grade 1 (=mild), Grade 2 (=moderate), Grade 3 (=severe) and Grade 4 (=potentially life-threatening).
Time Frame: Up to Day 12 post challenge
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Ad26.RSV.preF (1*10^11 vp) | Placebo
Number analyzed (Participants) | 27 | 26
Percentage of participants
  Heart rate: Abnormally low: Grade 1 | 0 | 3.8
  Heart rate: Abnormally low: Grade 2 | 0 | 3.8
  QTc Bazett (450 millisecond [ms], 480 ms) | 0 | 3.8
  QTc Bazett (increase from baseline [30; 60] ms) | 7.4 | 11.5
  QTc Fridericia: (increase from baseline [30; 60] ms) | 3.7 | 0

14. Secondary Outcome: Percentage of Participants With Clinical Laboratory Abnormalities (Graded)
Description: Percentage of participants with clinical laboratory abnormalities were reported. The biochemical and hematological parameters analyzed were- Alanine aminotransferase (AA), Alkaline phosphatase (AP), Aspartate aminotransferase (AsP), Hyperkalemia, Hypernatremia, Hypoglycemia, Hypophosphatemia, Hemoglobin, Neutrophils, White blood cell (WBC) - increase and Urine protein, which were graded by FDA Toxicity Grading Scale Grade 0 (=no grade), Grade 1 (=mild), Grade 2 (=moderate), Grade 3 (=severe) and Grade 4 (=potentially life-threatening).
Time Frame: Up to Day 28 post-challenge
Population: The Full Analysis Set (FAS) included all participants who were randomized and received at least one dose of study vaccine, regardless of the occurrence of protocol deviations. Here 'n' (number analyzed) signifies the number of participants analyzed for this OM at specified categories.
Measure: Number; unit: Percentage of participants
Arm/Group | Ad26.RSV.preF (1*10^11 vp) | Placebo
Number analyzed (Participants) | 31 | 32
Percentage of participants
  Post Dose: AA: Grade 1 | 9.7 | 0
  Post Dose: AP: Grade 1 | 0 | 3.1
  Post Dose: AsA: Grade 1 | 6.5 | 0
  Post Dose: AsA: Grade 2 | 0 | 3.1
  Post Dose: Hyperkalemia: Grade 2 | 3.2 | 0
  Post Dose: Hypernatremia: Grade 2 | 3.2 | 0
  Post Dose: Hypoglycemia: Grade 2 | 0 | 3.1
  Post Dose: Hypophosphatemia:Grade 1 | 3.2 | 0
  Post Dose: Hypophosphatemia:Grade 2 | 9.7 | 0
  Post Dose: Hemoglobin: Grade 1 | 3.2 | 3.1
  Post Dose: Hemoglobin: Grade 2 | 3.2 | 0
  Post Dose: Neutrophils: Grade 1 | 12.9 | 6.3
  Post Dose: WBC increase: Grade 1 | 0 | 3.1
  Post Dose: Urine Protein: Grade 1 | 3.2 | 3.1
  Post Challenge: AA: Grade 1: number analyzed (Participants) | 27 | 26
  Post Challenge: AA: Grade 1 | 25.9 | 15.4
  Post Challenge: AA: Grade 2: number analyzed (Participants) | 27 | 26
  Post Challenge: AA: Grade 2 | 7.4 | 3.8
  Post Challenge: AP: Grade 1: number analyzed (Participants) | 27 | 26
  Post Challenge: AP: Grade 1 | 0 | 3.8
  Post Challenge: AsA: Grade 1: number analyzed (Participants) | 27 | 26
  Post Challenge: AsA: Grade 1 | 14.8 | 15.4
  Post Challenge: AsA: Grade 2: number analyzed (Participants) | 27 | 26
  Post Challenge: AsA: Grade 2 | 3.7 | 3.8
  Post Challenge: AsA: Grade 4: number analyzed (Participants) | 27 | 26
  Post Challenge: AsA: Grade 4 | 0 | 3.8
  Post Challenge: Bilirubin: Grade 2: number analyzed (Participants) | 27 | 26
  Post Challenge: Bilirubin: Grade 2 | 3.7 | 0
  Post Challenge: Hyperglycemia: Grade 1: number analyzed (Participants) | 27 | 26
  Post Challenge: Hyperglycemia: Grade 1 | 0 | 3.8
  Post Challenge: Hyperkalemia: Grade 1: number analyzed (Participants) | 27 | 26
  Post Challenge: Hyperkalemia: Grade 1 | 3.7 | 3.8
  Post Challenge: Hypernatremia: Grade 2: number analyzed (Participants) | 27 | 26
  Post Challenge: Hypernatremia: Grade 2 | 3.7 | 0
  Post Challenge: Hypophosphatemia:Grade 1: number analyzed (Participants) | 27 | 26
  Post Challenge: Hypophosphatemia:Grade 1 | 3.7 | 0
  Post Challenge: Hypoproteinemia:Grade 1: number analyzed (Participants) | 27 | 26
  Post Challenge: Hypoproteinemia:Grade 1 | 11.1 | 0
  Post Challenge: Eosinophils: Grade 1: number analyzed (Participants) | 27 | 26
  Post Challenge: Eosinophils: Grade 1 | 0 | 7.7
  Post Challenge: Hemoglobin: Grade 1: number analyzed (Participants) | 27 | 26
  Post Challenge: Hemoglobin: Grade 1 | 7.4 | 0
  Post Challenge: Neutrophils: Grade 1: number analyzed (Participants) | 27 | 26
  Post Challenge: Neutrophils: Grade 1 | 7.4 | 0
  Post Challenge: Platelets: Grade 1: number analyzed (Participants) | 27 | 26
  Post Challenge: Platelets: Grade 1 | 3.7 | 3.8
  Post Challenge: Platelets: Grade 20: number analyzed (Participants) | 27 | 26
  Post Challenge: Platelets: Grade 20 | 0 | 3.8
  Post Challenge: WBC increase: Grade 1 | 3.7 | 0

ADVERSE EVENTS:
Time Frame: Up to 6 months post-vaccination and up to 6 months post-challenge
Description: The full analysis set (FAS) included all participants who were randomized and received at least one dose of study vaccine, regardless of the occurrence of protocol deviations.
Groups:
- Post-dose: Ad26.RSV.preF (1x10^11 vp): Participants received a single intramuscular injection of 1*10^11 vp (viral particles) of Ad26.RSV.preF on Day -28.
- Post-dose: Placebo: Participants received a single intramuscular injection of matching placebo on Day -28.
- Post-challenge: Challenge After Ad26.RSV.preF: Participants undergone intranasal challenge with RSV-A Memphis 37b virus on Day 0, after receiving single intramuscular doses of 1x1011 vp of Ad26.RSV.preF on Day -28.
- Post-challenge: Challenge After Placebo: Participants undergone intranasal challenge with RSV-A Memphis 37b virus on Day 0, after receiving single intramuscular doses of placebo on Day -28.
Arm/Group | Post-dose: Ad26.RSV.preF (1x10^11 vp) | Post-dose: Placebo | Post-challenge: Challenge After Ad26.RSV.preF | Post-challenge: Challenge After Placebo
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/32 | 0/27 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/32 | 1/27 | 0/26
Other Adverse Events (participants affected / at risk) | 4/31 | 9/32 | 16/27 | 16/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Post-dose: Ad26.RSV.preF (1x10^11 vp) (N=31) | Post-dose: Placebo (N=32) | Post-challenge: Challenge After Ad26.RSV.preF (N=27) | Post-challenge: Challenge After Placebo (N=26)
Ovarian Cyst (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Post-dose: Ad26.RSV.preF (1x10^11 vp) (N=31) | Post-dose: Placebo (N=32) | Post-challenge: Challenge After Ad26.RSV.preF (N=27) | Post-challenge: Challenge After Placebo (N=26)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 6 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Pharyngitis (Infections and infestations) | 0 | 0 | 3 | 4
Sunburn (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0
Alanine Aminotransferase Increased (Investigations) | 2 | 0 | 7 | 3
Aspartate Aminotransferase Increased (Investigations) | 2 | 1 | 2 | 2
Troponin T Increased (Investigations) | 0 | 0 | 0 | 2
Headache (Nervous system disorders) | 1 | 4 | 2 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 4
Dry Skin (Skin and subcutaneous tissue disorders) | 1 | 1 | 3 | 2

LIMITATIONS AND CAVEATS:
As no respiratory syncytial virus (RSV) vaccine has been previously tested in a human challenge model, the relationship between the results from this human challenge model and vaccine efficacy against natural infection is unknown.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation.

DOCUMENTS (2):
  • Study Protocol (2018-07-24): https://cdn.clinicaltrials.gov/large-docs/95/NCT03334695/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-30): https://cdn.clinicaltrials.gov/large-docs/95/NCT03334695/SAP_001.pdf